CLINICAL TRIAL: NCT06142123
Title: Comparative Effects Of 3-D Ankle Mobility Exercises And Eccentric Heel Drop Training In Female Athletes With Planter Fasciitis
Brief Title: Effects Of Ankle Mobility Exercises And Heel Drop Training In Planter Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0433
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Planter Fasciitis; Eccentric Heel Drop Training; 3-D Ankle Mobility
Keywords: Eccentric heel drop training, 3-D ankle mobility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will be treated with 3-D Ankle Mobility Exercises with combined isotonic (agonist) technique at ankle joint. Two diagonal (D2) Flexion-Extension patterns from the PNF leg patterns will be used.
  Both the techniques will be first performed in prone lying against the resistance of the therapist and then in crook lying.
  The patients will receive Intervention consisting 14 sets (7 sets for each 3-D extension-flexion [1 set (1 min) = exercise 30sec + rest 30 sec]) performed for 15 minutes thrice per week for four weeks
  Interventions: Other: 3-D Ankle Mobility Exercises(A)
- Group B (Experimental): Group B will be treated with Eccentric Heel Drop Training and Conventional physiotherapy treatment All patients will be treated once daily with 10 sets of 15 repetitions with a frequency of 2sec per repetitions and an interval of 30 sec between each set of Eccentric Heel drop training, 4 days a week for four weeks
  Interventions: Other: Eccentric Heel Drop Training(B)

INTERVENTIONS:
Other: 3-D Ankle Mobility Exercises(A) — The techniques will be first performed in prone lying against the resistance of the therapist and then in crook lying.
  1. The participant will perform the D2 extension pattern (Planter-flexion-supination inversion-toe flexion) using the CI technique in the prone position according to the resistance of therapist.
  2. The participant will perform the D2 flexion pattern (Dorsi-flexion-pronation eversion-toe extension) using CI technique in the prone position according to the resistance of therapist.
  3. The participant will perform the D2 extension pattern (Planter-flexion-supination inversion-toe flexion) using the CI technique in the crook-lying position according to the resistance of therapist.
  4. The participant will perform the D2 flexion pattern (Dorsi-flexion-pronation eversion-toe extension) using CI technique in the crook-lying position according to the resistance of therapist.
  Arms: Group A
Other: Eccentric Heel Drop Training(B) — : Group B will be treated with Eccentric Heel Drop Training. It will comprise of following exercises (14).
  1. Eccentric loading exercises of calf muscles.
  2. Conventional physiotherapy treatment including Ultrasound Plantar fascia stretching Calf muscle stretching Intrinsic muscles strengthening
  Arms: Group B

SUMMARY:
Planter fasciitis is a common cause of heel pain in adults. Planter fasciitis is frequently seen among athletes playing various sports. However, it is more prevalent in professional runner. The Biomechanical stresses including the increase in the intensity, frequency or the time frame of weight bearing activities that subject athlete's feet to continuous impact loads, surfaces with inadequate cushioning or improper shoe replacement are some of extrinsic risk factors associated with planter fasciitis.3-D ankle mobility exercises are improvised for treatment of plantar fasciitis, these comprise D2 diagonal PNF leg patterns, comprising of flexion-abduction-internal rotation and extension-adduction-external rotation. Heel drop exercise training is another useful intervention used for treating PF; the protocol consists transferring their body weight onto the forefoot of their dominant legs while slightly flexing their ankles. To get back to baseline, the non-dominant leg is given more weight, and the dominant leg's knee was remained fully extended to maintain higher gastrocnemius activation.

A Randomized clinical trial will be conducted at Pakistan Sports Board and Boston Physiotherapy Clinic Lahore through consecutive sampling technique on patients which will be allocated through opaque sealed enveloped into Group A and Group B. Group A will be treated with 3-D ankle mobility exercises and Group B will be treated with eccentric heel drop training. Outcome measures tools will be conducted through NPRS, Foot and Ankle Ability Measure (FAAM) and The VISA-A questionnaire: An index of the severity of Achilles tendinopathy after four weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

DETAILED DESCRIPTION:
Planter fasciitis is a common cause of heel pain in adults with a major incidence seen in women. Planter fasciitis is frequently seen among athletes playing various sports. However, it is more prevalent in professional runners(1). A list of intrinsic risk factors are associated with this condition which can be linked with individual's anatomy, physiology, their mobility & function or it can be linked with degenerative changes(2). The Biomechanical stresses including the increase in the intensity, frequency or the time frame of weight bearing activities that subject athlete's feet to continuous impact loads, surfaces with inadequate cushioning or improper shoe replacement are some of extrinsic risk factors associated with planter fasciitis(3). Individuals experiencing PF employ compensatory techniques to lessen pain experienced at the plantar fascia's origin(4). They assume antalgic gait pattern, increasing support on the lateral and anterior faces of the foot to reduce the amount of time their heels are in contact with the ground in return affecting upright posture within the base of support due to these compensations, which alter joint position perception and muscle activations resulting in static and dynamic imbalances(5).3-D ankle mobility exercises are improvised for treatment of plantar fasciitis, these comprise D2 diagonal PNF leg patterns, comprising of flexion-abduction-internal rotation and extension adduction-external rotation(6). To increase coordination, joint range of motion, muscular strength, and eccentric control associated with PF, these exercises can be paired with the combined isotonic (CI) approach. This allows the concentric, eccentric, and stabilizing contractions of agonists to be performed without relaxation(7). Heel drop exercise training is another useful intervention used for treating PF; the protocol consists transferring their body weight onto the forefoot of their dominant legs while slightly flexing their ankles. To get back to baseline, the non-dominant leg is given more weight, and the dominant leg's knee was remained fully extended to maintain higher gastrocnemius activation(8). The heel drop exercise modify Lateral and medial gastrocnemius architectural conditions which has been implicated in patients with PF, resulting in injury prevention(9).The purpose of our study is to determine a comparable exercise regime for planter fasciitis among athletes which can easily be incorporated as an essential component of their routine training program in order to prevent the occurrence of planter fasciitis as well as improve the prognosis of already affected athletes. Planter fasciitis is a common condition prevalent among female athletes, however, frequently ignored as well. The groundwork of this research will help creating awareness among female athletes and provide them with a significant solution to help with the pain which causes a less efficient exercise performance. Very few data is available to support the use of 3-d Ankle mobility exercises. Our investigation will also explore the generic effects of commonly unknown 3-d Ankle Mobility exercises with combined isotonic technique which are based on the D2 diagonal PNF patterns

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis based on the clinical presentation Pain on palpation along the proximal plantar fascia with or without radiographic evidence of a plantar calcaneal bone spur Pain reporting of minimum of 2 on NPRS Athletes with 18 years to 35 years of age Chronic plantar fasciitis of more than 3 months. Female athletes playing more than 2 years in sports including runners, Soccer players, cricket players, cyclist, body builders.

Exclusion Criteria:

Chronic pain syndrome or other foot pains Peripheral vascular disease that results in rest pain or intermittent claudication or venous stasis ulceration Calcaneal stress fracture or show evidence of a foreign body or tumor of the affected heel as viewed radio graphically Pregnant females Previously suffered a rupture or surgery of the plantar fascia within the 5 years preceding participation in the investigation Existing or prior osteomyelitis of the involved calcaneus

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female athletes
Enrollment: 26 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-05 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | pre and 4 weeks post interventional
  The Foot and Ankle Ability Measures Scale is a collection of self-administered questionnaire comprising 29 questions that is split down into two subscales: activities of daily living (21 questions) and sports population (8 questions)(15). With an ICC value of 0.89 for Activities of Daily Living (ADL) and 0.87 for the Sports subscale, it has a significant level of reliability
Numeric Pain Rating Scale | pre and 4 weeks post interventional
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10.
  0 indicates "no pain" and 10 indicates "worst pain"

SECONDARY OUTCOMES:
The VISA-A questionnaire: An index of the severity of Achilles tendinopathy: The VISA-A questionnaire: An index of the severity of Achilles tendinopathy | pre and 4 weeks post interventional
  The VISA-A is a self-administered questionnaire that aims to evaluate the clinical severity for patients with chronic Achilles tendinopathy and associated biomechanical abnormalities. It is an easily self-administered questionnaire that evaluates symptoms and their effect on physical activity. The three clinically significant patient-relevant domains of pain, function, and activity are assessed using the VISA-A questionnaire.
  In patients with AT, the VISA-A questionnaire exhibits strong test-retest reliability and has been validated (construct validity)

CONTACTS AND LOCATIONS:
Overall Officials: Muniba Afzal, Principal Investigator — Riphah International University
Locations (1):
- Boston Physiotherapy Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trojian T, Tucker AK. Plantar Fasciitis. Am Fam Physician. 2019 Jun 15;99(12):744-750. PMID 31194492
- [Background] Petraglia F, Ramazzina I, Costantino C. Plantar fasciitis in athletes: diagnostic and treatment strategies. A systematic review. Muscles Ligaments Tendons J. 2017 May 10;7(1):107-118. doi: 10.11138/mltj/2017.7.1.107. eCollection 2017 Jan-Mar. PMID 28717618
- [Background] Alonso-Fernandez D, Taboada-Iglesias Y, Garcia-Remeseiro T, Gutierrez-Sanchez A. Effects of the Functional Heel Drop Exercise on the Muscle Architecture of the Gastrocnemius. J Sport Rehabil. 2020 Nov 1;29(8):1053-1059. doi: 10.1123/jsr.2019-0150. Epub 2019 Dec 6. PMID 31810057
- [Background] Konrad A, Gad M, Tilp M. Effect of PNF stretching training on the properties of human muscle and tendon structures. Scand J Med Sci Sports. 2015 Jun;25(3):346-55. doi: 10.1111/sms.12228. Epub 2014 Apr 10. PMID 24716522
- [Background] Johannsen F, Olesen JL, Ohlenschlager TF, Lundgaard-Nielsen M, Cullum CK, Jakobsen AS, Rathleff MS, Magnusson PS, Kjaer M. Effect of Ultrasonography-Guided Corticosteroid Injection vs Placebo Added to Exercise Therapy for Achilles Tendinopathy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2219661. doi: 10.1001/jamanetworkopen.2022.19661. PMID 35816306